CLINICAL TRIAL: NCT07376109
Title: Effect of Infertility and Assisted Reproductive Technology (ART) on Sexual Function and Behaviour
Brief Title: Effects of Infertility and Assisted Reproductive Technology on Sexual Function and Behavior
Status: Not yet recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Michael Dahan, Assistant Professor, Department of Obstetrics and Gynecology; Reproductive Endocrinology and Infertility, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: MUHC-2025-11459
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Infertility Assisted Reproductive Technology; Sexual Behavior; Sexual Function; Sexual Dysfunction and Infertility; Sexual Dysfunction Female; Infertility; Assisted Reproductive Techniques
Keywords: infertility; Assisted Reproductive Technology; ART; IVF; female sexual function; female sexual function index; FSFI; sexual behavior; sexual dysfunction; women's sexual health
MeSH Terms: conditions — Sexual Behavior; Sexual Dysfunction, Physiological; Infertility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Infertility Cohort: Women attending the MUHC Reproductive Centre for evaluation or treatment of infertility who complete a single anonymous questionnaire assessing sexual function and sexual behaviour.

SUMMARY:
This cross-sectional observational study examines how infertility and the use of assisted reproductive technology (ART) are related to sexual function and sexual behaviors in women seeking fertility treatment. Infertility and the stress of ART may be associated with changes in sexual desire, satisfaction, and activity. The purpose is to better understand these associations to support the sexual health and overall well-being of women undergoing fertility care.

Women who are assigned female at birth, under 45 years old, diagnosed with infertility, and attending appointments at the MUHC Reproductive Centre are invited to take part. Participants will be asked to complete an anonymous questionnaire while waiting for their clinical visit. The questionnaire includes the validated Female Sexual Function Index (FSFI), which measures different aspects of sexual function, and additional questions about sexual activities, such as frequency of intercourse and other behaviors before and after fertility treatments.

Participants will not provide any identifying information. Completed questionnaires will be placed in a secure collection box to protect confidentiality.

Data from approximately 500 participants will be analyzed to explore how infertility type (primary vs. secondary), duration of infertility, and the number of unsuccessful ART cycles relate to sexual function and behavior. Findings from this study may help healthcare providers better recognize and address the sexual health concerns of women with infertility.

This study is approved by the McGill University Health Centre Research Ethics Board (REB #2025-11459).

DETAILED DESCRIPTION:
This is a single-center, cross-sectional observational study conducted at the McGill University Health Centre (MUHC) Reproductive Centre. The study is designed to examine associations between infertility characteristics and sexual function and sexual behaviors among women undergoing fertility treatment.

Participants are recruited in person during routine clinic visits. Anonymous, paper-based questionnaires are distributed by a research assistants. Questionnaires are completed voluntarily while participants are waiting for their appointment and returned anonymously into a secure collection box. No identifying information is collected at any time, and responses are not linked to medical records.

Sexual function is assessed using the validated Female Sexual Function Index (FSFI), which evaluates multiple domains of sexual function, including desire, arousal, lubrication, orgasm, satisfaction, and pain. Additional survey items assess sexual behaviors and changes in sexual activity patterns in the context of infertility and fertility treatment. Infertility-related variables include duration of infertility, type of infertility (primary vs. secondary), and history of fertility treatments, including unsuccessful treatment cycles.

Data from completed questionnaires are entered into a secure electronic database. Surveys that do not meet inclusion criteria based on self-reported responses are excluded from analysis.

The planned sample size is approximately 500 participants, based on clinic volume and feasibility over a 12-month recruitment period. This sample size is expected to provide sufficient power to detect clinically meaningful differences in sexual function scores across infertility subgroups.

Statistical analyses will include descriptive statistics to summarize participant characteristics, infertility variables, sexual function scores, and sexual behaviors. Comparisons between groups (e.g., primary vs. secondary infertility) will be performed using t-tests, and analyses across infertility duration categories will use analysis of variance (ANOVA). Pearson correlation coefficients will be used to examine relationships between the number of unsuccessful fertility treatment cycles and sexual function outcomes. Multivariable linear regression models will be constructed to evaluate the independent associations between infertility-related factors and sexual function while adjusting for relevant demographic variables. Missing data will be assessed for patterns and handled using appropriate statistical methods depending on the extent and nature of missingness.

Study data will be stored securely in accordance with institutional policies. Paper questionnaires are stored in locked cabinets, and electronic data are password-protected with restricted access. Data will be retained for five years following study completion and then securely destroyed. No future use of the data is planned.

ELIGIBILITY:
Inclusion Criteria:

1. Assigned female at birth.
2. Self-identify as a woman.
3. Age 18-44 years.
4. Diagnosis of infertility.
5. Seeking fertility treatment at the MUHC Reproductive Centre.

Exclusion Criteria:

1. Assigned male at birth.
2. Age 45 years or older.
3. Sexual practices that do not allow for the possibility of conception (e.g., same-sex relationships without use of assisted reproductive technologies).
4. Seeking oocyte cryopreservation.
5. Individuals who do not wish to complete the anonymous questionnaire.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All individuals who self-identify as women and were assigned female at birth are eligible to participate. Individuals assigned male at birth or who do not self-identify as women are excluded.
Study Population: This study will include women assigned female at birth, aged 18-44 years, who are seeking fertility treatment at the MUHC Reproductive Centre and have a diagnosis of infertility. Participants must self-identify as women. Individuals assigned male at birth, age 45 or older, seeking oocyte cryopreservation, or whose sexual practices do not allow for conception without assisted reproductive technologies will be excluded. Participation is voluntary and anonymous.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Female sexual function | Day 1
  Female sexual function as assessed using the validated Female Sexual Function Index (FSFI), which evaluates desire, arousal, lubrication, orgasm, satisfaction, and pain. Higher scores indicate better sexual function.
Sexual Behaviour | Day 1
  Self-reported sexual behaviors, including intercourse frequency (pre- and post-fertility treatment), oral sex, anal sex, masturbation, and other sexual practices, as assessed by the anonymous questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- MUHC Reproductive Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because all data are collected anonymously using paper questionnaires, contain no personal identifiers, and participants did not provide consent for data sharing beyond the scope of this study.